CLINICAL TRIAL: NCT03015246
Title: Biobehavioral Studies of Opioid Seeking: Effects of Buprenorphine/Naloxone Dose on Experimental Stress Reactivity and Opioid Abstinence
Brief Title: Effects of Buprenorphine/Naloxone Dose on Experimental Stress Reactivity and Opioid Abstinence
Acronym: BOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor of Psychiatry and Behavioral Neurosciences; and Director, Substance Abuse Research Division, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BOS-1
Record Dates: First submitted 2016-12-16; First posted 2017-01-10 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Heroin Dependence; Opioid Use Disorder
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Buprenorphine; Naloxone

STUDY DESIGN:
Intervention Model Description: 4x2 within-subject crossover design: 4 medication conditions (morphine first, then 3 doses of buprenorphine/naloxone), crossed with 2 stress conditions (placebo vs. stress [yohimbine + hydrocortisone], nested within medication conditions)
Who Masked: Participant, Outcomes Assessor
Masking Description: Medication conditions blinded using different-sized buprenorphine/naloxone sublingual tablets including placebo. Stress conditions blinded using encapsulation of yohimbine/placebo and hydrocortisone/placebo. Only pharmacy aware of drug codes.
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Extended-Release Morphine + placebo stressor (Placebo Comparator): Participants will be maintained on extended-release morphine (dose tailored to the individual, based on pre-experimental opioid use amount), in three divided daily doses. The placebo stressor will be administered on one day.
  Interventions: Drug: Extended release morphine; Drug: Placebo stressor
- Buprenorphine/Naloxone low dose + placebo stressor (Experimental): Participants will be maintained on Buprenorphine/Naloxone (Zubsolv™) sublingual tablet doses of 1.4/0.36 mg/day. The placebo stressor will be administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone low dose; Drug: Placebo stressor
- Buprenorphine/Naloxone moderate dose + placebo stressor (Experimental): Participants will be maintained on Buprenorphine/Naloxone (Zubsolv™) sublingual tablet doses of 4.2/1.08 mg/day. The placebo stressor will be administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone moderate dose; Drug: Placebo stressor
- Buprenorphine/Naloxone high dose + placebo stressor (Experimental): Participants will be maintained on Buprenorphine-Naloxone (Zubsolv™) sublingual tablet doses of 12.8/3.16 mg/day. The placebo stressor will be administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone high dose; Drug: Placebo stressor
- Extended-Release Morphine + active stressor (Experimental): Participants will be maintained on extended-release morphine (dose tailored to the individual, based on pre-experimental opioid use amount), in three divided daily doses. Yohimbine 60mg powder + Hydrocortisone (Cortef™) 20mg tablet administered on one day.
  Interventions: Drug: Extended release morphine; Drug: Active stressor
- Buprenorphine/Naloxone low dose + active stressor (Experimental): Participants will be maintained on Buprenorphine/Naloxone (Zubsolv™) sublingual tablet doses of 1.4/0.36 mg/day. The placebo stressor will be administered on one day. Yohimbine 60mg powder + Hydrocortisone (Cortef™) 20mg tablet administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone low dose; Drug: Active stressor
- Buprenorphine/Naloxone moderate dose + active stressor (Experimental): Participants will be maintained on Buprenorphine/Naloxone (Zubsolv™) sublingual tablet doses of 4.2/1.08 mg/day. Yohimbine 60mg powder + Hydrocortisone (Cortef™) 20mg tablet administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone moderate dose; Drug: Active stressor
- Buprenorphine/Naloxone high dose + active stressor (Experimental): Participants will be maintained on Buprenorphine-Naloxone (Zubsolv™) sublingual tablet doses of 12.8/3.16 mg/day. Yohimbine 60mg powder + Hydrocortisone (Cortef™) 20mg tablet administered on one day.
  Interventions: Drug: Buprenorphine/Naloxone high dose; Drug: Active stressor

INTERVENTIONS:
Drug: Extended release morphine — Dose (tailored to each participant based on his/her pre-experimental opioid use amount) is administered in 3 divided daily doses.
  Arms: Extended-Release Morphine + active stressor; Extended-Release Morphine + placebo stressor
Drug: Buprenorphine/Naloxone low dose — Buprenorphine/Naloxone dose of 1.4/0.36 mg/day
  Other Names: Zubsolv™ sublingual tablet
  Arms: Buprenorphine/Naloxone low dose + active stressor; Buprenorphine/Naloxone low dose + placebo stressor
Drug: Buprenorphine/Naloxone moderate dose — Buprenorphine/Naloxone dose of 4.2/1.08 mg/day
  Other Names: Zubsolv™ sublingual tablet
  Arms: Buprenorphine/Naloxone moderate dose + active stressor; Buprenorphine/Naloxone moderate dose + placebo stressor
Drug: Buprenorphine/Naloxone high dose — Buprenorphine/Naloxone dose of 12.8/3.16 mg/day
  Other Names: Zubsolv™ sublingual tablet
  Arms: Buprenorphine/Naloxone high dose + active stressor; Buprenorphine/Naloxone high dose + placebo stressor
Drug: Active stressor — Yohimbine hydrochloride 60mg + Hydrocortisone 20mg tablet
  Arms: Buprenorphine/Naloxone high dose + active stressor; Buprenorphine/Naloxone low dose + active stressor; Buprenorphine/Naloxone moderate dose + active stressor; Extended-Release Morphine + active stressor
Drug: Placebo stressor — Lactose
  Arms: Buprenorphine/Naloxone high dose + placebo stressor; Buprenorphine/Naloxone low dose + placebo stressor; Buprenorphine/Naloxone moderate dose + placebo stressor; Extended-Release Morphine + placebo stressor

SUMMARY:
This research deals with behaviors that are part of opioid dependence. The purpose is to study how stress and medication dose can affect opioid drug use.

DETAILED DESCRIPTION:
If participants meet all the criteria, their involvement in the study (Phases 1 and 2 described below) will last for 10-13 weeks. Participants will be asked to stay at the research site for a minimum of 2 nights on 4 separate weeks and will have 22 office visits During that time, participants can't leave the unit unescorted or have visitors.

Participants will receive a medication called Buprenorphine/Naloxone. Buprenorphine/Naloxone is approved by the Food and Drug Administration (FDA) to treat opioid addiction, and is a safe and effective alternative to methadone. Participants will receive this medication every day. When participants are not living on the inpatient unit they will come to the research clinic every day to receive the medication.

On Day 1, one single 1-mL (0.2 teaspoon) blood sample will be collected to assess the effect of the Buprenorphine/Naloxone medication dose on gene expression pattern.

On each day of admission (once on weeks 3, 5 and 7), a single 1-mL (0.2 teaspoon) blood sample will be collected to assess the effect of the buprenorphine/naloxone medication dose on the participant's gene expression pattern.

On the 8 days while participants are an inpatient they will participate in experimental sessions that involve drug administration. On some days participants will receive morphine and on some days participants will receive oral medications called yohimbine and hydrocortisone that will be used to study stress responses. Each afternoon study staff will collect one blood sample (10 mL or 2 teaspoons) from a vein in the participant's arm; these samples will be used to measure biological signals of stress.

At the end of the study participants will be detoxified from the Buprenorphine/Naloxone medication over a 3-week outpatient period.

Study participants will be scheduled for one separate in-person visit at 1 month after week 11. At this follow-up visit participants will be asked to provide a urine sample and to complete questionnaires that ask about drug craving and use, withdrawal symptoms, risky situations for drug use, coping with stress, and consequences experienced from using drugs or being abstinent.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent, as determined by structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Willing to use an adequate form of contraception for the duration of the study.
* Reads and writes English
* Participants must be in generally good health to be eligible. All candidates will receive a routine medical exam (history and physical) with standard laboratory tests (including blood and urine samples, EKG, mandatory TB testing, and voluntary HIV testing).

Exclusion Criteria:

* No candidate who has a current DSM-IV Axis I disorder other than Drug Dependence or a history of serious psychiatric problems (e.g. psychosis, bipolar or major depression) will be allowed to participate.
* Candidates meeting criteria for opioid or nicotine dependence will not be excluded, but those with other Substance Dependence disorders will be excluded. Those with Abuse of Alcohol, Cannabis, Cocaine, will not be excluded, but participants must provide an alcohol free breath specimen.
* No candidate with medical (neurological, cardiovascular, pulmonary or systemic) disorders will be allowed to participate. This will be determined with history and physical exam, standard laboratory testing (blood and urine), EKG, and TB tests (to avoid transmitting this communicable disease on the residential unit or in the laboratory).
* Candidates with evidence of cognitive impairment (based on reading ability and comprehension, will be excluded.
* Female candidates who are pregnant (urine pregnancy test), lactating, or not using adequate birth control methods (self-report) will be excluded.
* Candidates with injection phobia, or seeking treatment for opioid dependence will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Opioid price-inelasticity (economic demand) | measured once (end of session) in each of the 8 experimental sessions over 7 weeks
  demand intensity (L) and demand elasticity (a) on hypothetical drug purchasing task

SECONDARY OUTCOMES:
Opioid Symptom Questionnaire: Agonist symptoms | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  Total opioid agonist symptom score (16 items, each scored on 0-4 scale, for a scale score range of 0-64, with higher scores indicating higher opioid agonist symptoms)
Opioid Symptom Questionnaire: Withdrawal symptoms | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  Total opioid withdrawal symptom score (16 items, each scored on 0-4 scale, for a scale score range of 0-64, with higher scores indicating higher withdrawal symptoms)
Visual Analog Scale (VAS) ratings | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  VAS ratings will measure "liking", "good drug effect," "bad drug effect," "stimulated," "sedated", "[preferred opioid] craving", and "cigarette craving". Each VAS is scored from 0 (not at all) to 100 (extremely).
Profile of Mood States (POMS) | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  72-item POMS questionnaire, which has several subscale scores
Blood pressure | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  Systolic/diastolic blood pressure (mm Hg)
Heart rate | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  Heart rate (beats/min)
Pupil diameter | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline 0930, 1030, 1145, 1230, 1300, 1330, 1400, 1430, 1500, and 1600.
  Pupil diameter (mm) measured with digital pupillometer
Plasma noradrenaline level | Measured once per session at 2-hours post Yohimbine in each of the 8 experimental sessions
  Plasma noradrenaline level (µg/ml)
Plasma BDNF level (µg/ml) | Measured once per session at 2-hours post Yohimbine in each of the 8 experimental sessions
  Plasma brain derived neurotrophic factor level (pg/ml)
Plasma IL-1Ra level (µg/ml) | Measured once per session at 2-hours post Yohimbine in each of the 8 experimental sessions
  Plasma interleukin 1Ra level (pg/ml)
Saliva cortisol level | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline, 1.5, 2, 3 and 4 hours post Yohimbine in each of the 8 experimental sessions.
  Saliva cortisol level (µg/dL)
Saliva alpha-amylase level | Within-session change is being assessed, in each of 8 sessions over 7 weeks. Within-session measurements at baseline, 1.5, 2, 3 and 4 hours post Yohimbine in each of the 8 experimental sessions.
  Saliva alpha-amylase level (U/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Vince and Associates, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No